CLINICAL TRIAL: NCT03952949
Title: A Default Option to Enhance Dietary Quality in Participants With Food Insecurity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University at Albany (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 16-E-260-01
Record Dates: First submitted 2019-05-14; First posted 2019-05-16 (Actual); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Nutrition Poor
Keywords: Nutrition; Food Insecurity; Choice Architecture; Nudge
MeSH Terms: conditions — Malnutrition | interventions — Nutrition Assessment

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Default (Experimental): Participants in the default condition were presented with a pre-filled online shopping cart containing a combination of groceries that meet macro- and micronutrient requirements for their gender and age, and told that they are free to delete, add, and exchange any item they wish to finalize their selections.
  Interventions: Behavioral: Default Option While Online Grocery Shopping
- Nutrition Education (Active Comparator): Participants in the nutrition education condition were instructed to read a brief education brochure before online grocery shopping.
  Interventions: Behavioral: Nutrition Education

INTERVENTIONS:
Behavioral: Default Option While Online Grocery Shopping — The "default option" is a behavioral economics construct that refers to the option a consumer selects if no active choice is made (e.g. opt-out 401K plans, which significantly increase enrollment, compared to active sign up). Participants in the default condition were presented with a prefilled online shopping cart containing groceries that met nutritional requirements based on participants' gender and age.
  Arms: Default
Behavioral: Nutrition Education — The nutrition education materials were adapted from materials currently utilized by the New York State Office of Temporary and Disability Assistance ("Eat Smart New York").
  Arms: Nutrition Education

SUMMARY:
Food insecurity is associated with an increased risk of overweight/obesity and weight-related chronic illnesses. The availability of a default option (i.e., option a consumer selects if no active choice is made) has been shown to effectively nudge consumer behavior. An online default option (i.e., prefilled grocery shopping cart) was previously shown to positively impact food selection in an online grocery shopping task.The present study provides preliminary evidence for the efficacy of an online default option in enhancing the nutritional quality of online grocery purchases in individuals with food insecurity.

DETAILED DESCRIPTION:
Food insecurity is associated with an increased risk of overweight/obesity and weight-related chronic illnesses. The present study provides preliminary evidence for the efficacy of an online default option in enhancing the nutritional quality of online grocery purchases in individuals with food insecurity.

In behavioral economics, the default option refers to the option a consumer selects if no active choice is made. This study aims to determine whether the use of a default prefilled online grocery shopping cart results in the purchase of healthier food items in individuals with food insecurity, compared to nutrition education. The default approach, a non-monetary intervention that manipulates choice architecture, improves food choice behaviors in individuals facing significant financial constraints. The intervention is potentially broadly scalable via online platforms.

It was hypothesized that the default option effectively increases the nutritional quality of foods purchased online, compared to nutrition education.

Fifty participants recruited from food pantries in New York in 2018 were randomized to: (1) review nutrition information before selecting groceries for a week using a local grocery store's online shopping and delivery service (n = 23) or (2) modify a default prefilled online shopping cart containing groceries that meet nutritional guidelines according to their personal preferences (n = 27).

Primary outcome measures capture the nutritional quality of groceries purchased. Our primary nutritional outcomes include servings of whole grains fruits and vegetables, fiber, daily calories, fat, saturated fat, sodium and cholesterol content.

ELIGIBILITY:
Inclusion Criteria:

1. age 18 or older
2. single person household
3. fluent in written and spoken English
4. able to provide informed consent
5. food-insecure (verbal agreement that they consider themselves to be of that category) but not currently receiving SNAP benefits (as they would otherwise have access to twice the amount of benefits typically allocated; please note that all participants will be provided with information about enrollment in SNAP following study participation)
6. current residence in a zip code served by Price Chopper's delivery program

Exclusion Criteria:

1. None of the following dietary restrictions: vegetarian/vegan, gluten-free/celiacs disease, and lactose intolerant
2. current residence outside of a zip code served by Price Chopper's delivery program

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-01-04 (Actual); Primary Completion 2017-10-28 (Actual); Study Completion 2017-10-28 (Actual)

PRIMARY OUTCOMES:
Nutritional Quality of Groceries Purchased | Single visit, <1.5 hours
  The Thrifty Food Plan Calculator (TFPC) was used to quantify the nutritional quality of groceries selected by study participants. The TFPC was developed using U.S. Department of Agriculture nutrition and consumption data and is designed to have users input information about the relative amount of money spent on various categories of food and provides comprehensive information on caloric, macro-, and micronutrient content of the foods selected based on participant age and gender.

CONTACTS AND LOCATIONS:
Overall Officials: Julia M. Hormes, PhD, Principal Investigator — University at Albany

IPD SHARING:
Plan to Share IPD: No